CLINICAL TRIAL: NCT03723538
Title: Efficacy and Safety of Dexmedetomidine Sedation in Spontaneous Breathing Patients After Tracheal Surgery
Brief Title: Dexmedetomidine Use for Sedation in Patients Submitted to Tracheal Surgery
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Silvia Fiorelli, principal investigator, University of Roma La Sapienza
Other Study IDs: DEX=!
Record Dates: First submitted 2018-10-18; First posted 2018-10-29 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Dexmedetomidine — patients undergoing tracheal resection and reconstruction surgery were enrolled in this prospective observational pilot study to evaluate dexmedetomidine-based sedation after tracheal surgery in an Intensive Care Unit (ICU). Patients remain electively intubated with an uncuffed nasal endotracheal tube, awake and exhibit spontaneous breathing The neck was maintained in flexion through chin-to-chest sutures. Infusion of dexmedetomidine was started from a dosage of 0.7 μg kg-1 h-1 followed by dose titration to the target level of the sedation Richmond Agitation Sedation Scale, (RASS) score -1/-2 using a dose range of 0.2-1.4 μg kg-1 h-1.

SUMMARY:
Patients undergoing tracheal resection and reconstruction surgery are enrolled in this prospective observational pilot study to evaluate dexmedetomidine-based sedation after tracheal surgery in an Intensive Care Unit (ICU). Patients remain electively intubated with an uncuffed nasal endotracheal tube, awake and exhibit spontaneous breathing The neck was maintained in flexion through chin-to-chest sutures. Infusion of dexmedetomidine was started from a dosage of 0.7 μg kg-1 h-1 followed by dose titration to the target level of the sedation Richmond Agitation Sedation Scale, (RASS) score -1/-2 using a dose range of 0.2-1.4 μg kg-1 h-1.

ELIGIBILITY:
Inclusion Criteria:

* patients submitted to tracheal surgery
* elective surgery
* age ≥ 18 years

Exclusion Criteria:

* severe neurological disorder
* visual or hearing impairment
* acute cerebrovascular disease
* mean arterial pressure (MAP) <55 mmHg or hypotension requiring the use of inotropes/vasopressors
* heart rate (HR) <50 bpm
* second and third degree atrioventricular block (AV block) in the absence of PMK
* Sequential Organ Failure Assessment (SOFA) score <2 index
* hepatic failure
* emergency surgery
* pregnancy
* patient refusal to give consent
* inability to give consent
* age ≤18 years
* ASA score ≥ IV.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective tracheal resection and reconstruction surgery and admitted to ICU after surgery
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the efficacy in changing the sedation level during the infusion | at T0 (baseline) and 12 hours from the beginning of the infusion
  monitored through the sedation scale called Richmond Agitation-Sedation Scale(RASS).RASS is a medical scale used to measure the agitation or sedation level of a person.The score ranges from +4 "combative" to -5 "unarousable". The target level of the sedation is a RASS score -1/-2 .

SECONDARY OUTCOMES:
The secondary endpoint is evaluation of safety throughout the incidence of adverse effects during the infusion | at T0 (baseline), 3, 6, 12 and 18 hours from the beginning of the infusion)
  by recording modification of MAP, HR, and SpO2. Any cardiorespiratory complications (hypotension with MAP<60 mmHg or 50% baseline reduction, bradycardia with HR <40 bpm or reduction of greater than 50% of the baseline value, and desaturation with SpO2 <90%) were also recorded.pain control assessed by VAS, need of rescue doses of alternative drugs

CONTACTS AND LOCATIONS:
Locations (1):
- azienda ospedaliero universitaria Sant'Andrea, Roma, Italy

IPD SHARING:
Plan to Share IPD: No